CLINICAL TRIAL: NCT02998736
Title: PERIOP-04 Phase Ib Trial of Perioperative Tadalafil and Influenza Vaccination in Cancer Patients Undergoing Major Surgical Resection of a Primary Abdominal Malignancy
Brief Title: Trial of Perioperative Tadalafil and Influenza Vaccination in Cancer Patients Undergoing Major Surgical Resection of a Primary Abdominal Malignancy
Acronym: PERIOP-04
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20160855-01H
Record Dates: First submitted 2016-12-06; First posted 2016-12-20 (Estimated); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Abdominal Cancer
Keywords: Colon
MeSH Terms: interventions — Tadalafil; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Cialis 20 mg daily by mouth for 16 day. 5 days prior to surgery, day of surgery and 10 days post surgery.
  Influenza vaccine 0.5mL day of surgery
  Interventions: Drug: Cialis; Biological: Influenza vaccine
- Control (No Intervention): No intervention in the perioperative period

INTERVENTIONS:
Drug: Cialis — Cialis 20 mg daily by mouth for 16 day. 5 days prior to surgery, day of surgery and 10 days post surgery.
  Influenza vaccine 0.5mL day of surgery
  Other Names: Tadalafil
  Arms: Intervention
Biological: Influenza vaccine — One 0.5mL intramuscular injection the day of surgery
  Other Names: Agriflu
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine if giving Cialis for 5 days prior to surgery, on the day of surgery along with the influenza vaccine and Cialis 10 days after surgery will have an affect at the cell level for decreasing the chances of the spread of disease post surgery.

DETAILED DESCRIPTION:
Surgical resection of a primary malignancy, while critical for cure, results in postoperative immune suppression, characterized by MDSC mediated inhibition of NK cell killing. In preclinical models the causal link between this immune suppression and the formation of postoperative metastases is undeniable. Fortunately, this postoperative immune suppression is preventable using modulators of MDSC and NK cell function. In this Phase Ib study the hypothesis is that simultaneous administration of perioperative tadalafil, to prevent MDSCs from suppressing NK cells, and influenza vaccine, to directly activate NK cells will safely and effectively reverse the effects of surgical stress on NK cell cytotoxicity. This is a necessary first step towards demonstrating that this re-purposed perioperative regimen can reduce the formation of postoperative metastatic disease in cancer surgery patients.

In this proposed Phase I trial a carefully selected promising perioperative immunomodulatory regimen, which includes tadalafil and influenza vaccination, for rapid clinical translation. The proposal is to re-purpose these drugs, they already have ample safety data associated with their use but neither agent has been systematically administered immediately prior to surgery. This trial will allow us to not only establish the safety of this regimen but will permit a rigorous assessment of its ability to reverse surgery-induced suppression of NK cells. If this regimen can effectively prevent postoperative NK cell dysfunction without any regimen limiting toxicity then this will provide the necessary data required to undertake a randomized efficacy study in a specific cancer subtype, with cancer recurrence as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of a primary abdominal malignancy consented to undergo major surgery with a planned length of stay of 3 or more days.
* Eligible patients must have signed a consent for surgical resection of the malignancy.
* Adequate hematological function defined as: platelet count ≥ 100 x 109/L, absolute neutrophil count ≥ 1 x 109/L, white blood count ≥ 2.5 x 109/L, hemoglobin count ≥ 90 g/L.
* Adequate organ functioning, including: total bilirubin ≤ 1.5 x upper limit of normal (ULN); AST, ALT < 2.5 x ULN; INR <1.5 ; CrCl>30mL/min.
* If sexually active, and of childbearing potential, subjects must agree to use acceptable birth control from screening until the final study visit (study day, SD35) or early termination. Acceptable methods of birth control include: spermicide with condom, diaphragm, or cervical cap, IUD (intrauterine device), hormonal contraception, vasectomy, and abstinence. (Plan B or the rhythm method are not considered reliable methods.
* Male subjects should agree to avoid having sex for 5 days before surgery and 10 days post surgery taking tadalafil due to the risk of sustained erection
* Ability to understand and provide a signed informed consent form (ICF) approved by the Institutional Review Board (IRB/IEC/REB).
* Ability to comply with protocol requirements.

Exclusion Criteria:

* Prior adjuvant chemotherapy or radiation within 8 weeks of planned surgery.
* Pregnant or nursing mothers or women of childbearing potential not using acceptable methods of birth control.
* Documented significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication (e.g. systemic corticosteroids, azathioprine, cyclosporin A). Subjects may be on physiologic doses of replacement prednisone or equivalent doses of corticosteroid (<7.5 mg daily).
* History of autoimmune disease (even if controlled with medication) such as but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis.
* Allergies or any contraindication to the use of tadalafil or any components of Cialis® or the influenza vaccine (including eggs), Agriflu®.
* Serious intercurrent chronic or acute illness, or other illness considered by the investigator as an unwarranted high risk for an investigational product.
* Patients who have suffered a myocardial infarction, stroke, or life-threatening arrhythmia within the last 6 months.
* Patients with resting hypotension (BP <90/50 at rest) or hypertension (BP >170/110 at rest).
* Patients with cardiac failure or coronary artery disease causing unstable angina.
* Use any type of nitrate drug therapy, including short-acting nitrate-containing medications, due to the risk of developing potentially life-threatening hypotension. The use of organic nitrates, either regularly and/or intermittently, in any form (e.g. oral, sublingual, transdermal, by inhalation) is absolutely contraindicated (see list Appendix II).
* Use of guanylate cyclase stimulators (cinaciguat or riociguat).
* Use of alpha-blocker therapy (see list in Appendix I).
* Previous episode of non-arteritic anterior ischaemic optic neuropathy (NAION) or history of retinitis pigmentosa.
* Use of anti-platelet (excluding ASA) or anti-coagulation medication (Patients who discontinue such medications at least 7 days prior to first treatment may be eligible for this study).
* Use of the following anti-viral agents: ribavirin, adefovir, cidofovir (at least 7 days prior to the first treatment), and PEG-IFN (at least14 days prior to the first treatment).
* Active infection of any site requiring ongoing treatment.
* Known anatomical deformities of the penis (such as angulation, cavernosal fibrosis or Peyronie's disease) or any condition that might predispose the patient to priapism.
* History of Guillaine-Barré Syndrome.
* Subjects with a medical or psychological impediment to probable compliance with the protocol should be excluded.
* Active drug or alcohol use or dependence or other conditions that, in the opinion of the investigator, would interfere with adherence to study requirements. Social alcohol use is acceptable.
* Concurrent inhibitors of moderate or strong CYP3A4 inhibitors
* Taking any other PDE-5 inhibitor (such as sildenafil) during the active phase of the study between enrollment to SD35.
* History of lactose or milk sugar intolerance
* Liver or Kidney disease
* Sickle cell anemia
* Peptic ulcer or other bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Determine the change in the number of regimen limiting toxicities (RLT) in the experimental cohort | measured at day 1, 3, 7, 10 and 35 post surgery
  Adverse events, vitals and medications will be collected.
Document the change in the number and severity of CTCAE adverse events that are probably or definitely related to study treatment (tadalafil or influenza) in the experimental cohort. | measured at day 1, 3, 7, 10 and 35 post surgery
  Adverse events reported

SECONDARY OUTCOMES:
Compare the reduction in Natural Killer cell killing as measured on PBMC collected on SD1 as compared to baseline between the control and experimental cohorts, using a standard Natural Killer cell killing assay (51Chromium release assay). | measured on day 1, 3, 7, 10 and 35 post surgery blood specimens

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Auer, Doctor, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hirsch C, Zorger AM, Baumann M, Park YS, Brockelmann PJ, Mellinghoff S, Monsef I, Skoetz N, Kreuzberger N. Vaccines for preventing infections in adults with solid tumours. Cochrane Database Syst Rev. 2025 Apr 16;4(4):CD015551. doi: 10.1002/14651858.CD015551.pub2. PMID 40237463